CLINICAL TRIAL: NCT01363791
Title: Effect of Fructose on Metabolic Control in Humans: A Series of Systematic Reviews and Meta-analyses to Provide Evidence-based Guidance for Nutrition Guidelines Development
Brief Title: Meta-analyses of Fructose and Cardiometabolic Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Calorie Control Council (Other)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Adjunct Research Fellow, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CIHR-KS-2009-205030
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia; Diabetes; Prediabetes; Dysglycemia; Overweight; Obesity; Gout; Hypertension; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; High fructose corn syrup; Fruit; Isocaloric; Hypercaloric; Cardiometabolic risk factors; Triglycerides; Cholesterol; Glycemic control; Insulin resistance; Body weight; Uric acid; Blood pressure; Fatty liver; Fasting; Postprandial
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus; Prediabetic State; Overweight; Obesity; Gout; Hypertension; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Cardiovascular Diseases; Insulin Resistance; Body Weight; Fatty Liver; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dietary fructose — Oral dietary fructose in free (unbound) form in isocaloric exchange for other non-fructose carbohydrate sources (isocaloric trials) or added to a control diet as a source of excess energy (hypercaloric trials).

SUMMARY:
Diabetes and heart associations continue to discourage high intakes of dietary fructose, a constituent part of the sucrose molecule that is found in fruits and vegetables as a natural sugar and in some processed foods and beverages as an added sweetener. The concern relates to its ability to increase certain blood fats and cholesterol, which increase the risk of cardiovascular disease. The evidence for an adverse effect of fructose on these risk factors, however, is inconclusive. To improve the evidence on which nutrition recommendations for fructose are based, the investigators therefore propose to study the effect of fructose on blood fats, cholesterol, sugars, blood pressure, and body weight, by undertaking a systematic synthesis of the data taken from all available clinical studies in humans. This technique has the strength of allowing all of the available data to be pooled together and differences to be explored in groups of different study participants (healthy humans of different sex, weight, and age and in those with diseases which predispose to disturbances in metabolism, such as diabetes) with dietary fructose in different forms, doses, and with differing durations of exposure. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing recommendations for the general public, as well as those at risk of diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
Background: Fructose has been implicated in chronic disease guidelines. The American Heart Association (AHA) and American (ADA), Canadian (CDA), and European (EASD) Diabetes Associations discourage dietary fructose at high intakes (>15-20% energy), citing its ability to aggravate blood lipids. The American Heart Association (AHA) and the World Health Organization (WHO) recommend reduced consumption (<5-7% and <10% energy, respectively) of added sugars, especially as high fructose corn syrup in sugar sweetened beverages, to decrease the risk of weight gain. These concerns, however, are based on inconsistent intervention data in humans. There is also paradoxical evidence that small, catalytic doses of fructose at a level obtainable from fruit (<10-g/meal) may improve glycemic control in humans.

Objective: To improve evidence-based guidance for fructose recommendations, the investigators propose conducting a series of 7 systematic reviews and meta-analyses of controlled feeding trials to assess the effect of oral fructose on cardiometabolic risk in humans. The first 6 systematic reviews and meta-analyses will each be conducted on a different area of cardiometabolic risk: (1) lipids, (2) glycemic control, (3) body weight, (4) uric acid, (5) blood pressure, and (6) non-alcoholic fatty liver (NAFL). The seventh meta-analysis will investigate the effect of small, "catalytic" doses of fructose at a level obtainable from fruit (<10-g/meal) on all areas of cardiometabolic risk.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources. MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms, supplemented by manual, hand searches of bibliographies.

Study selection: We will include controlled feeding trials investigating the effect of fructose in isocaloric exchange for other carbohydrate sources (isocaloric trials) or added to a control diet as a source of excess energy (hypercaloric trials) on cardiometabolic risk factors in humans. Studies that are <7-days diet duration, lack a control, or do not provide viable endpoint data will be excluded. To isolate the effects of fructose, we will also exclude trials in which fructose was administered exclusively as sucrose (bound fructose) or high-fructose corn syrup (42% to 55% of free fructose), except where these sweeteners were the comparator.

Data extraction. Two investigators will independently extract information about study design, sample size, subject characteristics, fructose form, dose, reference-carbohydrate, follow-up, and background diet profile. Mean±SEM values will be extracted for all outcomes. Standard computations and imputations will be used to derive missing variance data. Investigators will assess the quality/validity of each study using the Heyland Methodological Quality Score (MQS).

Outcomes: The first 6 of 7 proposed analyses will each assess a set of outcomes related to a different area of cardiometabolic risk: (1) lipids (fasting lipids [triglycerides, HDL-cholesterol [C], LDL-C, apo-B, total-C:HDL-C ratio, apo-B:apo-A1 ratio, non-HDL-C] and postprandial lipids(non-fasting peak, mean, and area under the curve [AUC] triglycerides), (2) glycemic control (fasting glucose and insulin, glycated blood proteins) and insulin sensitivity (Euglycemic-hyperinsulinemic clamp, frequent sampling intravenous glucose tolerance test [FSIGT], Homeostasis model assessment of insulin resistance [HOMA-IR], oral glucose tolerance test insulin sensitivity index [OGTT-ISI]), (3) body weight, (4) uric acid, (5) blood pressure (systolic BP, diastolic BP, mean arterial pressure), and (6) NAFL (imaging and spectroscopy endpoints of liver fat and biomarkers of hepatocellular injury [transaminases]). The last proposed analysis investigating the effect of small, "catalytic" doses of fructose will focus on all 6 outcomes.

Data synthesis. Meta-analyses will be conducted using the Generic Inverse Variance method applying random effects models expressed as standardized mean differences (SMDs) with 95% CIs. Paired analyses will be applied for crossover trials according to Elbourne et al. (Int J Epidemiol. 2002;31:140-149). Heterogeneity will be assessed by the Q statistic and quantified by I2. A priori subgroup analyses will be undertaken to explore sources of heterogeneity including the effect of underlying disease status, reference carbohydrate (comparator), fructose form, dose, follow-up, study design, baseline measurements, and study quality on the effect of fructose. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, level of feeding control, energy balance and composition of the background diet, etc.) and sensitivity analyses. Meta-regression analyses will assess the significance of subgroups analyses with piece-wise meta-regression techniques used to identify dose or follow-up thresholds. Publication bias will be investigated by inspection of funnel plots.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Preliminary findings: A pilot project which explored the effect of fructose on lipids in diabetes identified 786 articles, of which 14 (16 trials)were included in a meta-analysis. Isocaloric exchange of fructose for carbohydrate had a triglyceride raising effect in type 2 diabetes only where the reference carbohydrate was starch, dose was >60-g/d, or follow-up was ≤4-weeks. These distinctions had not been appreciated previously (Sievenpiper et al. Diabetes Care 2009;32:1930-1937).

Significance: The proposed project will aid in knowledge translation related to the effects of dietary fructose on diabetes, and cardiovascular risk factors, strengthening the evidence-base for recommendations and improving health outcomes through informing consumers and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Trials in humans
* Oral fructose intervention
* Suitable control (i.e. another carbohydrate source in isocaloric exchange for fructose or a control diet which is compared with the same diet supplemented with excess energy from fructose)
* >= 7-days diet duration
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* IV or parenteral fructose
* High fructose corn syrup or sucrose intervention (except where these are the comparators)
* Lack of a suitable control
* < 7-days diet duration.
* No viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Varied.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Lipid Analysis | June 2012
  Analyses:
  1. Fasting lipids (triglycerides, HDL-cholesterol [C], LDL-C, apo-B, total-C:HDL-C ratio, apo-B:apo-A1 ratio, non-HDL-C)
  2. Postprandial lipids (peak, mean, and area under the curve [AUC] triglycerides)
Body Weight Analysis | November 2011
  Analyses:
  1. Body weight
Glycemic Control Analysis | June 2012
  Analyses:
  1. Glycated blood proteins (HbA1c, fructosamine, glycated albumin), glucose, and insulin in people with diabetes
  2. Glycated blood proteins (HbA1c, fructosamine, glycated albumin), glucose, and insulin in people without diabetes
  3. Insulin sensitivity (Euglycemic-hyperinsulinemic clamp, frequent sampling intravenous glucose tolerance test [FSIGT], Homeostasis model assessment of insulin resistance [HOMA-IR], oral glucose tolerance test insulin sensitivity index [OGTT-ISI])
Blood Pressure (BP) Analysis | January 2012
  Analyses:
  1. Systolic BP, diastolic BP, and mean arterial pressure (MAP)
Uric Acid Analysis | February 2012
  Analyses:
  1. uric acid
"Catalytic" Fructose Across Cardiometabolic Endpoints Analysis | January 2012
  Analyses:
  1. Lipids, glycemic control, body weight, blood pressure, and uric acid
Non-Alcoholic Fatty Liver (NAFL) Analysis | June 2012
  Analyses:
  1. Imaging and spectroscopy endpoints of liver fat (Liver ultrasound [US], computed tomography [CT], magnetic resonance imaging [MRI], or magnetic resonance spectroscopy [MRS]) and biomarkers of hepatocellular injury (transaminases [ALT, AST, GGT])

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Study Director — Department of Pathology and Molecular Medicine, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Micheal's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, Carleton AJ, Chatha S, Jiang HY, de Souza RJ, Beyene J, Kendall CW, Jenkins DJ. Heterogeneous effects of fructose on blood lipids in individuals with type 2 diabetes: systematic review and meta-analysis of experimental trials in humans. Diabetes Care. 2009 Oct;32(10):1930-7. doi: 10.2337/dc09-0619. Epub 2009 Jul 10. PMID 19592634
- [Result] Ha V, Sievenpiper JL, de Souza RJ, Chiavaroli L, Wang DD, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Dibuono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Hypertension. 2012 Apr;59(4):787-95. doi: 10.1161/HYPERTENSIONAHA.111.182311. Epub 2012 Feb 13. PMID 22331380
- [Result] Sievenpiper JL, de Souza RJ, Mirrahimi A, Yu ME, Carleton AJ, Beyene J, Chiavaroli L, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. Effect of fructose on body weight in controlled feeding trials: a systematic review and meta-analysis. Ann Intern Med. 2012 Feb 21;156(4):291-304. doi: 10.7326/0003-4819-156-4-201202210-00007. PMID 22351714
- [Result] Wang DD, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. The effects of fructose intake on serum uric acid vary among controlled dietary trials. J Nutr. 2012 May;142(5):916-23. doi: 10.3945/jn.111.151951. Epub 2012 Mar 28. PMID 22457397
- [Result] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Result] Sievenpiper JL, de Souza RJ, Jenkins DJ. Sugar: fruit fructose is still healthy. Nature. 2012 Feb 22;482(7386):470. doi: 10.1038/482470e. No abstract available. PMID 22358823
- [Result] Sievenpiper JL, de Souza RJ, Kendall CW, Jenkins DJ. Is fructose a story of mice but not men? J Am Diet Assoc. 2011 Feb;111(2):219-20; author reply 220-2. doi: 10.1016/j.jada.2010.12.001. No abstract available. PMID 21272692
- [Result] David Wang D, Sievenpiper JL, de Souza RJ, Cozma AI, Chiavaroli L, Ha V, Mirrahimi A, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on postprandial triglycerides: a systematic review and meta-analysis of controlled feeding trials. Atherosclerosis. 2014 Jan;232(1):125-33. doi: 10.1016/j.atherosclerosis.2013.10.019. Epub 2013 Nov 2. PMID 24401226
- [Result] Sievenpiper JL, de Souza RJ, Cozma AI, Chiavaroli L, Ha V, Mirrahimi A. Fructose vs. glucose and metabolism: do the metabolic differences matter? Curr Opin Lipidol. 2014 Feb;25(1):8-19. doi: 10.1097/MOL.0000000000000042. PMID 24370846
- [Result] Sievenpiper JL; Toronto 3D (Diet, Digestive Tract, and Disease) Knowledge Synthesis and Clinical Trials Unit. Fructose: where does the truth lie? J Am Coll Nutr. 2012 Jun;31(3):149-51. doi: 10.1080/07315724.2012.10720021. No abstract available. PMID 23204150
- [Result] Chiavaroli L, Ha V, de Souza RJ, Kendall CW, Sievenpiper JL. Re. "Association of fructose consumption and components of metabolic syndrome in human studies: a systematic review and meta-analysis". Nutrition. 2015 Feb;31(2):419-20. doi: 10.1016/j.nut.2014.07.018. Epub 2014 Aug 8. No abstract available. PMID 25441580
- [Derived] Chiavaroli L, de Souza RJ, Ha V, Cozma AI, Mirrahimi A, Wang DD, Yu M, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ, Sievenpiper JL. Effect of Fructose on Established Lipid Targets: A Systematic Review and Meta-Analysis of Controlled Feeding Trials. J Am Heart Assoc. 2015 Sep 10;4(9):e001700. doi: 10.1161/JAHA.114.001700. PMID 26358358
- [Derived] Cozma AI, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Wang DD, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on glycemic control in diabetes: a systematic review and meta-analysis of controlled feeding trials. Diabetes Care. 2012 Jul;35(7):1611-20. doi: 10.2337/dc12-0073. PMID 22723585